CLINICAL TRIAL: NCT02269163
Title: A Phase 3, Multicenter, Open-Label Study of the Safety, Tolerability, Efficacy, and PK of ProMetic BioTherapeutics IGIV (Human) 10% in Adults and Children With Primary Immunodeficiency Diseases
Brief Title: Study of ProMetic BioTherapeutics Immune Globulin Intravenous (Human) 10%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prometic Biotherapeutics, Inc. (Industry)
Collaborators: Atlantic Research Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2004C009G
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gammargard, Gammaplex, Gamunex, or Octogam Treatment Period (Active Comparator): Subjects who enroll in the study while on Gammargard, Gammaplex, Gamunex, or Octogam IGIV Product and need to wait for the scheduled start of Prometic IGIV (10%) treatment will continue on their usual dose and treatment cycle with Gammargard, Gammaplex, Gamunex, or Octogam IVIG Product during this period.
  Interventions: Biological: Immune Globulin Intravenous
- Prometic IGIV 10% Treatment Period (Experimental): Subjects will receive Prometic Immune Globulin Intravenous 10%
  Interventions: Biological: Prometic's Immune Globulin Intravenous 10%

INTERVENTIONS:
Biological: Immune Globulin Intravenous — Gammargard, Gammaplex,Gamunex, or Octogam IGIV Product
  Arms: Gammargard, Gammaplex, Gamunex, or Octogam Treatment Period
Biological: Prometic's Immune Globulin Intravenous 10% — Liquid formulation of Prometic Immune Globulin Intravenous 10% (human) in 50 mL vials containing 100 mg/mL of immunoglobulin G (IgG)
  Arms: Prometic IGIV 10% Treatment Period

SUMMARY:
Phase 3 multicenter, open-label study of safety, tolerability, efficacy, and pharmacokinetics (PK) of ProMetic's Immune Globulin Intravenous (Human) 10%, the investigational medicinal product [IMP]), in Adults and Children with Primary Immunodeficiency Diseases (PIDD).

DETAILED DESCRIPTION:
This is a pivotal Phase 3, open-label, single-arm, multicenter study to assess the tolerability, safety, efficacy, and Pharmacokinetics of the Investigational Medicinal Product in adults and children with Primary Immunodeficiency Diseases (PIDD). A total of approximately 75 subjects aged 2-80 years will be enrolled in the study. Subjects who switch from an investigational immune globulin or subcutaneous immune globulin (IGSC) are required to receive a stable dose of commercial product (CP), which is a licensed commercially available immune globulin intravenous (IGIV) product for at least 3 cycles before they can be given the Investigational Medicinal Product . This study schema will result in the Commercial Product Treatment Period and Investigational Medicinal Product Treatment Period. All subjects will be treated on an outpatient basis with the Investigational Medicinal Product for approximately 1 year, with the dose and schedule based on their previous IGIV treatment regimen (21-day or 28-day dosing interval). A subset of subjects will participate in a Pharmacokinetics sub-study.

The primary objective of the study is to examine the rate of clinically documented serious bacterial infections (SBIs) in subjects treated with the Investigational Medicinal Product to achieve a rate of less than one SBI per year.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between the ages of 2 and 80 years at Screening.
2. Female subjects of childbearing potential must agree to employ adequate birth control measures, as determined by their IRB/IEC, for the duration of the study.
3. The subject must have one of the following three diagnoses (isolated PIDD of other types will be excluded):

   * Common variable immunodeficiency
   * X-linked agammaglobulinemia
   * Hyper-IgM syndrome and documented low IgG levels (<4.5 mg/mL [450 mg/dL]).
4. Subjects must have been treated with a stable dose of immune globulin administered intravenously (IGIV) or subcutaneously (IGSC) and has documented trough or steady state IgG levels of ≥ 5 mg/mL.

Exclusion Criteria:

1. Subject has secondary immunodeficiency or has been diagnosed with dysgammaglobulinemia or isolated IgG subclass deficiency; has known hypoalbuminemia (<3 gm/dL), protein-losing enteropathy, or nephrotic syndrome.
2. Subject has ever had a history of severe anaphylactic or anaphylactoid reaction to immunoglobulins or other blood products.
3. Subject has a known history of immunoglobulin A (IgA) deficiency and known anti-IgA antibodies, thrombotic event, such as deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism, at any time.
4. Subject has received blood products except IGIV, IGSC, or albumin within the previous 12 months or has participated in another study (except for IGIV, IGSC studies) within the previous 4 weeks.
5. Subject has had cancer in the past 5 years, except for basal cell or squamous cell cancers of the skin.
6. Subject has had a documented active infection within 7 days prior to Screening, or subject is on continuous prophylactic antibiotics.
7. Subject is positive for human immunodeficiency virus (HIV)-1 or HIV-2, a positive hepatitis C virus (HCV) or hepatitis B virus (HBV).
8. Subject has levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 times the upper limit of normal (ULN).
9. Subject has serum creatinine >1.5 times the ULN or a severe chronic condition such as renal failure with proteinuria.
10. Subject has anemia with a hemoglobin level ≤8 g/dL.
11. Subject has severe neutropenia with neutrophil count ≤1000 per mmᴧ3 or has lymphopenia with <500 per/ mmᴧ3.
12. Subject is taking prednisone at a dose ≥0.15 mg/kg/day and receiving other immunosuppressive drugs or chemotherapy.
13. Subject has known atrial fibrillation requiring anticoagulant therapy; congestive heart failure (New York Heart Association Class III/IV); cardiomyopathy; or cardiac arrhythmia associated with thromboembolic events, unstable or advanced ischemic heart disease, or hyperviscosity.
14. Subject has known decreased Protein C and/or Protein S levels.
15. Subject is positive for antibodies to β2GPI and/or β2GPI DI at Screening.
16. Female subject who is pregnant, breast-feeding, or planning a pregnancy during the course of the study.
17. A history of epilepsy or multiple episodes of migraine (defined as at least one episode within 6 months of enrolment) not completely controlled by medication, or any condition that is likely to interfere with evaluation of the IMP or satisfactory conduct of the study in the Investigator's opinion.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Moy, MD, Study Chair — Rush University Medical Center
Locations (13):
- United States (13):
  - University of California, Irvine, Irvine, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Immunoe International Research, Centennial, Colorado
  - National Jewish Hospital, Denver, Colorado
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Fort Wayne Medical Institute, Fort Wayne, Indiana
  - St. Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Optimed Research, Columbus, Ohio
  - Dallas Allergy Immunology, Dallas, Texas
  - Bellingham Asthma, Allergy and Immunology Clinic, Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The term "Participants" for the overall study period reflects the number of subjects included in the analysis of the Prometic IGIV 10% Treatment period (75 subjects).
Groups:
- Cohort 1 - Adult: The Prometic IGIV 10% Treatment Period was the elapsed time from the first administration of Prometic IGIV 10% to study completion. Cohort 1 consisted of adult subjects aged 17-80 years.
- Cohort 2 - Pediatric: The Prometic IGIV 10% Treatment Period was the elapsed time from the first administration of Prometic IGIV 10% to study completion. Cohort 2 consisted of pediatric subjects aged 2 to < 17 years.
Period: Overall Study
Arm/Group | Cohort 1 - Adult | Cohort 2 - Pediatric
Started | 50 | 25
Completed | 47 | 18
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Major protocol violation | 0 | 1
Not completed — Other | 2 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Adult | Cohort 2 - Pediatric | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Median (Full Range); unit: years] | 57 [17 to 75] | 9 [3 to 15] | 42.0 [3 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 5 | 36
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 45 | 19 | 64
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 46 | 24 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Time since first Primary Immune Deficiency Disease (PIDD) diagnosis (years) [Median (Full Range); unit: years] | 12 [0.9 to 39.5] | 1.9 [0.3 to 14.1] | 6.4 [0.3 to 39.5]

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Occurrence of Serious Bacterial Infections (SBI)
Description: SBIs were calculated for each subject as 52n/w, where n is the number of reported SBIs and w is the number of weeks on study. For the combined cohorts only, a 99% one-sided (upper) confidence limit for the incidence rate of SBIs (scaled to represent 12 months exposure if necessary) was derived, and the objective of demonstrating that the true infection rate was below 1 per subject per year was considered established if this upper limit was less than 1. To calculate the confidence limit, a negative binomial regression model will be used. This model includes an overdispersion parameter to account for possible intra-subject correlation as well as the actual time period each subject is on the study as an offset variable.
Time Frame: One year
Population: CP Treatment Period and Prometic IGIV 10% Treatment Period: Analysis was performed on the all treated population, which consisted of all subjects who are enrolled into the study and received study treatment (CP or Prometic IGIV 10%) Prometic IGIV 10% Treatment Period Cohort 1 and Cohort 2: Analysis was performed on the all treated population, which consisted of all subjects who are enrolled into the study and received study treatment
Measure: Number (99% Confidence Interval); unit: Rate of events per subject per year
Groups:
- CP Treatment Period: The CP Treatment Period was the elapsed time from enrollment to the first administration of Prometic IGIV 10%; this was also known as the CP Waiting Period. During this time period, subjects received either their current CP or a CP chosen by the Investigator in consultation with their treating physician.
- Prometic IGIV 10% Treatment Period: The Prometic IGIV 10% Treatment Period was the elapsed time from the first administration of Prometic IGIV 10% to study completion
- Prometic IGIV 10% Treatment Period (Cohort 1): The Prometic IGIV 10% Treatment Period was the elapsed time from the first administration of Prometic IGIV 10% to study completion (adult population)
- Prometic IGIV 10% Treatment Period (Cohort 2): The Prometic IGIV 10% Treatment Period was the elapsed time from the first administration of Prometic IGIV 10% to study completion (pediatric population)
Arm/Group | CP Treatment Period | Prometic IGIV 10% Treatment Period | Prometic IGIV 10% Treatment Period (Cohort 1) | Prometic IGIV 10% Treatment Period (Cohort 2)
Number analyzed (Participants) | 66 | 75 | 50 | 25
Rate of events per subject per year | 0 [NA to NA] — No SBIs detected | 0.01 [NA to 0.03] — No lower limit was calculated | 0 [NA to NA] — 1-sided 99% CI calculated for combined cohorts only | 0.03 [NA to NA] — 1-sided 99% CI calculated for combined cohorts only

2. Secondary Outcome: Trough Levels of IgG (Total) Prior to Each Prometic IGIV 10% Infusion
Description: Subject's total IgG levels will be assessed prior to each Prometic IGIV 10% infusion
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP Treatment Period | Prometic IGIV 10% Treatment Period | Prometic IGIV 10% Treatment Period (Cohort 1) | Prometic IGIV 10% Treatment Period (Cohort 2)
Number analyzed (Participants) | 66 | 75 | 50 | 25
mg/dL | 1075.131 (210.7547) | 1043.401 (208.3044) | 1070.725 (219.3308) | 988.752 (175.7991)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were captured from the signing of informed consent/assent to 21 ± 4 days or 28 ± 4 days following the last infusion of study drug, an average of approximately 1 year per participant.
Description: Treatment-emergent adverse events (TEAEs) are presented for the safety population which consisted of all subjects who were enrolled into the study and recceived study product (Prometic IGIV 10% or CP). At each visit, AEs were elicited using a standard non-leading question such as "How have you been since the last visit / during the previous study period?" AEs were also elicited through the use of Subject Diary cards that the Investigator reviewed in detail with the subject at each visit
Arm/Group | CP Treatment Period | Prometic IGIV 10% Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/75
Serious Adverse Events (participants affected / at risk) | 5/66 | 7/75
Other Adverse Events (participants affected / at risk) | 57/66 | 72/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP Treatment Period (N=66) | Prometic IGIV 10% Treatment Period (N=75)
Bacteremia (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
False positive investigation result (Investigations) | 0 | 1
Adrenalectomy (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP Treatment Period (N=66) | Prometic IGIV 10% Treatment Period (N=75)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 9
Nausea (Gastrointestinal disorders) | 1 | 8
Vomiting (Gastrointestinal disorders) | 0 | 8
Chest pain (General disorders) | 0 | 4
Fatigue (General disorders) | 3 | 17
Local swelling (General disorders) | 1 | 4
Pain (General disorders) | 3 | 4
Pyrexia (General disorders) | 3 | 16
Acute sinusitis (Infections and infestations) | 3 | 10
Bronchitis (Infections and infestations) | 4 | 6
Conjunctivitis (Infections and infestations) | 1 | 4
Ear infection (Infections and infestations) | 2 | 7
Gastroenteritis viral (Infections and infestations) | 1 | 6
Influenza (Infections and infestations) | 3 | 6
Nasopharyngitis (Infections and infestations) | 4 | 8
Pharyngitis (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 14 | 16
Upper respiratory tract infection (Infections and infestations) | 13 | 18
Urinary tract infection (Infections and infestations) | 1 | 8
Viral upper respiratory tract infection (Infections and infestations) | 4 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 6
Procedural headache (Injury, poisoning and procedural complications) | 2 | 8
Procedural pain (Injury, poisoning and procedural complications) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 12
Dizziness (Nervous system disorders) | 5 | 7
Headache (Nervous system disorders) | 11 | 24
Migraine (Nervous system disorders) | 2 | 5
Paraesthesia (Nervous system disorders) | 1 | 4
Sinus headache (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 4 | 0
Haemosiderinuria (Renal and urinary disorders) | 5 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of data generated in the study is governed by the Investigator Clinical Trial Agreement

DOCUMENTS (2):
  • Study Protocol (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT02269163/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT02269163/SAP_001.pdf